CLINICAL TRIAL: NCT00910832
Title: Comparative, Randomized, Double-blind Study of the Efficacy of Eductyl® Versus Placebo for Treatment of Patients With Dyschesia Treated by Rectal Rehabilitation
Brief Title: Efficacy of Eductyl® Versus Placebo for Treatment of Dyschesia
Acronym: Eductyl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Techni Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-EDU-01; EudraCT N° : 2007-0003658-27
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Dyschesia
Keywords: Dyschesia treatment; Rehabilitation; Dyschesia
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eductyl suppository (Experimental)
  Interventions: Drug: Eductyl suppository
- Placebo suppository (Placebo Comparator)
  Interventions: Drug: Placebo suppository

INTERVENTIONS:
Drug: Eductyl suppository — one suppository every morning during 21 days
  Arms: Eductyl suppository
Drug: Placebo suppository — placebo suppository every morning during 21 days
  Arms: Placebo suppository

SUMMARY:
The purpose of this study is to assess the efficacy of Eductyl versus placebo for treatment of patients with dyschesia treated by rectal rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years
* Patients with dyschesia
* Prescription of rehabilitation for dyschesia

Exclusion Criteria:

* Rectal diseases
* Pain killers
* Pregnant women
* Breast feeding patients
* Non-compliant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of Eductyl versus placebo for treatment of patients with dyschesia treated by rectal rehabilitation on VAS of intensity of symptoms | Day -7, 0, 3, 7, 10, 14, 17, and 21

SECONDARY OUTCOMES:
To assess the efficacy on change symptoms and safety of Eductyl versus placebo for treatment of patients with dyschesia treated by rectal rehabilitation | Day 0 and 21

CONTACTS AND LOCATIONS:
Overall Officials: Odile Cotelle, Dr, Principal Investigator — Diaconesses hospital
Locations (1):
- Diaconesses Hospital, Paris, France

REFERENCES:
- [Derived] Cotelle O, Cargill G, Marty MM, Bueno L, Cappelletti MC, Colangeli-Hagege H, Savarieau B, Ducrotte P. A concomitant treatment by CO2-releasing suppositories improves the results of anorectal biofeedback training in patients with dyschezia: results of a randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2014 Jun;57(6):781-9. doi: 10.1097/DCR.0000000000000098. PMID 24807604